CLINICAL TRIAL: NCT01705496
Title: Sensitivity and Specificity of [124I]FIAU PET-CT Scanning in Patients Presenting With Pain in a Prosthetic Knee or Hip Joint
Brief Title: [124I]FIAU PET-CT Scanning in Patients With Pain in a Prosthetic Knee or Hip Joint
Acronym: PJI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sensitivity and specificity were not able to be assessed in this study due to the poor image quality.
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BVD002
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Prosthetic Joint Infections
Keywords: Phase II; FIAU; Fialuridine; Prosthetic; Joint; Infection; PET-CT
MeSH Terms: conditions — Infections | interventions — fialuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [124I]FIAU (Experimental): Single dose study of [124I]FIAU in patients presenting with pain in a prosthetic knee or hip joint who will undergo PET-CT scanning.
  Interventions: Radiation: [124I]FIAU

INTERVENTIONS:
Radiation: [124I]FIAU — This is a single dose study of 5 mCi [124I]FIAU in subjects presenting with pain in a prosthetic knee or hip joint. Subject will receive two PET-CT scans after [124I]FIAU injection.
  Other Names: Fialuridine

SUMMARY:
This protocol will evaluate the sensitivity and specificity of [124I]FIAU as a diagnostic imaging agent for the detection of prosthetic joint infections in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age >18 years
2. Ability to provide informed consent
3. A plain anterior-posterior (AP) and frog leg lateral X-ray of the hip or knee within 6 weeks of enrollment
4. Need for operative intervention in the opinion of the surgeon to correct the pain in the prosthetic joint
5. Prosthetic joint implant that has been in site for more than 3 months prior to enrolment
6. Having adequate general health to be expected to tolerate surgery adn to survive for 6 months from the time of informed consent
7. Women must be either postmenopausal or surgically sterile
8. Ability to return for all study assessments
9. Clinically euthyroid, or on stable thyroid replacement therapy

Exclusion Criteria:

1. Subjects who are unable to comply with study requirements
2. Indication, in the opinion of the principal investigator, for urgent surgery that would preclude the time needed for PET-CT scanning
3. History of an inherited mitochondrial disorder (e.g., Leber's hereditary neuropathy; neuropathy; ataxia, retinitis pigmentosa and ptosis [NARP]; myoneurogenic gastrointestinal encephalopathy [MNGIE]; myocolonic epilepsy with ragged red fibers [MERFF]; and mitochondrial myopathy, encephalomyopathy, lactic acidosis and stroke-like syndrome [MELAS])
4. Alanine aminotransferase (ALT) >5x the upper limit of normal (ULN) OR aspartate aminotransferase (AST) >5X ULN
5. Creatinine clearance <30 mL/min
6. Body mass that exceeds the rating of the CT table
7. Hypersensitivity to iodine
8. Any condition that would put the subject at reasonable risk in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Gulfcoast Research Institute, LLC, Sarasota, Florida
  - Phoenix Clinical Research, LLC, Tamarac, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Mission Hospital, Asheville, North Carolina
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Hosptial of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Trials of Texas, Incorporated, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | [124I]FIAU
Started | 23
Completed | 19
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Estimate the Sensitivity and Specificity of [124I]FIAU
Description: The sensitivity and specificity of [124I]FIAU in the detection of prosthetic joint infection was determined based on the correlation of the patient's infection status determined by an independent image reviewer and the infection status assessed by an adjudication committee.
  * Presence or absence of infection: Images were to be assessed and optimized on an ongoing basis. The single blinded reader was to assess independently the PET-CT images (attenuation corrected [AC] and non-AC PET plus the AC CT) and provide a diagnosis (infected or uninfected) using the chosen parameter(s) without knowing the results of the surgery. The radiology reviewer was not given any additional clinical information on the patient for reassessments relative to the initial reads. A separate central radiologist was to read the comparator X-rays independently for the presence or absence of infection. All pathology slides were to be read by a single pathologist. Local microbiology results were to be used.
Time Frame: 30 hours
Population: Out of 23 enrolled, only 22 received the investigational drug. One subject withdrew.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 22
percentage of participants | 80 [65 to 95]

2. Secondary Outcome: Evaluate the Safety and Tolerability of [124I]FIAU
Description: Safety will be monitored throughout the study for all subjects. safety will be assessed by monitoring of adverse events,vital signs,physical exams, and clinical laboratory tests including CBC, serum chemistry.
Time Frame: 30 +/- 2 days
Population: 22 received the investigational drug. A single IV injection of 5 mCi [124I]FIAU was well tolerated in patients presenting with pain in a prosthetic joint.
Measure: Number; unit: participants with adverse events
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 22
participants with adverse events | 15

3. Secondary Outcome: Define PET-CT Interpretation Criteria That Best Differentiate Infected vs Non-infected Prosthetic Joints
Description: The efficacy of [124I]FIAU could not be established due to the non-specific nature of the PET-CT signals caused by the metal artifacts from the prosthesis and pronounced muscle uptake of FIAU. It was impossible to define image review parameters for diagnosis of prosthetic joint infection.
Time Frame: 30 +/- 2 days
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 0

4. Secondary Outcome: Understand the Prevalence of Prosthetic Joint Infection
Description: The trial failed primary outcome, and this secondary outcome was not analyzed
Time Frame: 30 +/- 2 days
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Explore Whether the Adjudication Committee Evaluation of a Subject's Infection Status Correlates With Either of the Two Proposed Published Standards
Description: An independent adjudication committee will assess the totality of clinical information from each subject and assign them a status of infected or uninfected. The subject's infection status will be compared with either of the two proposed published standards to determine whether it corelates with any of the current consensus definitions or diagnostic algorithms.
  The trial failed primary outcome, and this secondary outcome was not analyzed.
Time Frame: 30 +/- 2 days
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Estimate the Sensitivity and Specificity of Plain X-ray in Detecting Prosthetic Joint Infection
Description: The adjudication committee evaluation of a subject's infection status will be used as the standard of truth to which X-ray is compared.
  The trial failed primary outcome, and this secondary outcome was not analyzed.
Time Frame: 15 mins
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Determine the Sensitivity and Specificity of [124I]FIAU vs. Plain X-ray in Detecting Prosthetic Joint Infection
Description: The adjudication committee evaluation of a subject's infection status will be used as the standard of truth to which [124I]FIAU and X-ray are compared.
  The trial failed primary outcome, and this secondary outcome was not analyzed.
Time Frame: 30 hours
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | [124I]FIAU
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 15/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [124I]FIAU (N=22)
Hypersensitivity to a concomitant drug (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [124I]FIAU (N=22)
Diarrhoea and nausea (Gastrointestinal disorders) | 4
Leukocytosis & Thrombocytosis (Blood and lymphatic system disorders) | 2
Injection site pain (General disorders) | 1
Urinary tract infection (Infections and infestations) | 2
procedural complications (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 1
Drug hypersensitivity (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days